CLINICAL TRIAL: NCT00741559
Title: Combined Role of PET and MEG in Nonlesional Epilepsy in Pediatric Population
Brief Title: Combined Role of Position Emission Tomography (PET) and Magnetoencephalography (MEG) in Nonlesional Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Amer Shammas, Nuclear Medicine Radiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000011429
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Epilepsy
Keywords: epilepsy; pediatrics; magnetoencephalography; electroencephalography; positron emission tomography
MeSH Terms: conditions — Epilepsy | interventions — Magnetoencephalography; Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: magnetoencephalography; Device: Positron emission tomography (PET); Device: Magnetic resonance imaging

INTERVENTIONS:
Device: magnetoencephalography — MEG studies are performed using a whole-head Omega 151-channel gradiometer system.
Device: Positron emission tomography (PET) — An interictal FDG(fluoro-D-glucose)-PET will be obtained in a single 10 minute scanning session. PET scans will be obtained using a 3D acquisition technique, which will allow the use of a lower dose of radiotracer.
Device: Magnetic resonance imaging — MR will be performed on a 1.5T or 3T system, using a combination of different sequences including sagittal T1, coronal and axial T2, FLAIR and proton density and axial 3D T1 weighted images.

SUMMARY:
The first aim of this study are to evaluate the lobar concordance of FDG-PET and MEG with intracranial electrographic study in children with intractable partial epilepsy. The second aim is to determine if the combined role of FDG-PET and MEG improve detection of epileptogenic zone as defined by invasive intracranial recordings.

DETAILED DESCRIPTION:
Children with poorly controlled epilepsy are extensively investigated with various tools including MR brain, electroencephalography (EEG), magnetoencephalography (MEG) or position emission tomography (PET) scans. When MR brain does not show an abnormality, the patient is said to have nonlesional epilepsy. In these cases, it is even more crucial to be able to identify the epileptogenic zone, depending on availability of investigative tool.

Recognizing that individual modalities have limitations, the aim of this study is to determine if combining non-invasive investigations with MEG and PET, which respectively evaluate the electrical and metabolic activity of the brain, could improve the children with intractable nonlesional epilepsy with MEG and PET and compared this with invasive intracranial monitoring. The endpoint of the study being agreement on localizations of epileptogenic zone using PET and MEG individually and in combination and comparing this with invasive intracranial monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages 0-18 years with (1) nonlesional intractable focal epilepsy and (2) those with discordant clinical and EEG findings, who are potential surgical candidates

Exclusion Criteria:

* Patients who are pregnant

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The concordance rate of FDG-PET and MEG with video EEG | 3 years

SECONDARY OUTCOMES:
The positive and negative predictive values of each modality and combined modalities in assessing the epileptogenic zone. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Charron, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada